CLINICAL TRIAL: NCT00110734
Title: A Randomized, Double-Blind, Placebo Controlled, Paired Study Evaluating S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) for Induction of Local Dermal Anesthesia for Laser-Assisted Tattoo Removal in Adults
Brief Title: S-Caine™ Peel (Skin Numbing Cream) to Treat Pain During Laser-Assisted Tattoo Removal in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: SCP-43-05
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%)

SUMMARY:
There is pain associated with laser-assisted tattoo removal. For this reason, some form of anesthesia is commonly used to eliminate or minimize the pain. This anesthesia is usually a topical local anesthetic cream or ointment spread over the skin. The purpose of this study is to further estimate the effectiveness of S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) for treating pain during laser-assisted tattoo removal.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient elects to undergo laser-assisted tattoo removal

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient has participated in a clinical trial of an unapproved drug within the previous 30 days
* Patient has participated in any previous clinical trial involving S-Caine Peel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2005-09

PRIMARY OUTCOMES:
To evaluate the efficacy of S-Caine Peel when applied for 60 minutes for induction of local dermal anesthesia prior to laser-assisted tattoo removal in adults

SECONDARY OUTCOMES:
To monitor the nature and frequency of adverse events (AEs) associated with the application of S-Caine Peel

CONTACTS AND LOCATIONS:
Locations (1):
- Laser and Skin Surgery Center of New York, New York, New York, United States